CLINICAL TRIAL: NCT05048082
Title: A Phase 2, Single-Dose, Open-Label Study to Evaluate Diagnostic Performance and Safety of Pegsitacianine, an Intraoperative Fluorescence Imaging Agent for the Detection of Lung Malignancies, in Patients Undergoing Routine Surgery
Brief Title: A Study to Evaluate Pegsitacianine, an Intraoperative Fluorescence Imaging Agent for the Detection of Lung Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoNano Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ON-1005
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: An interventional, open-label, single arm trial where each patient is his/her own intrapatient control. All patients will receive a single dose of pegsitacianine administered intravenously prior to standard of care (SOC) surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluorescence imaging with pegsitacianine (Experimental): Pegsitacianine 1 mg/ml infused 24-72 hours prior to surgery.
  Interventions: Drug: pegsitacianine; Procedure: Tumor resection surgery

INTERVENTIONS:
Drug: pegsitacianine — An intraoperative nanoparticle-based fluorescence imaging agent comprised of micelles covalently conjugated to indocyanine green (ICG).
  Other Names: ONM-100
Procedure: Tumor resection surgery — Standard of care surgical removal of cancerous lung lesion

SUMMARY:
This Phase 2 study is an open-label, single-arm trial where each patient is his/her own "intrapatient" control. All patients will receive a single dose of pegsitacianine prior to standard of care surgery.

DETAILED DESCRIPTION:
This single-arm trial will enroll patients with biopsy confirmed or a high clinical suspicion of a lung malignancy based on MRI, CT and/or PET imaging. A total of up to 40 patients will be enrolled in this trial. The sponsor reserves the right to perform an interim analysis following early enrollment (i.e., n ≤ 10 subjects) to determine the feasibility and benefit of pegsitacianine as an adjunct to standard of care surgical resection of lung malignancies.

The surgeon will begin by attempting to perform their SOC tumor resection. If the tumor is unable to be located under standard white light conditions, an appropriate FDA-cleared near-infrared imaging device may be used to aid in the location of the primary tumor. Localization of the primary tumor, when unable to be located using white light imaging, in conjunction with pathology confirmed presence of disease will be considered a clinically significant event. Following any standard of care procedures conducted under white light only, the near infrared camera will be used to evaluate areas of residual fluorescence that may be resected if suscpicious for metastatic spread or residual margins. The fluorescence status of each specimen will then be correlated to the final pathology for each, and performance metrics of pegsitacianine will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis, or a high clinical suspicion of a lung malignancy based on MRI, CT and/or PET imaging

Exclusion Criteria:

* Known hypersensitivity or allergy to indocyanine green (ICG), polymethylmethacrylate (PMMA; found in dental and bone cements) or polyethylene glycol (PEG)
* Tumor locations the surgeon deems unfeasible to image intraoperatively
* Excessive and/or generalized disease deemed inoperable by the surgeon
* Life expectancy less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — Penn Medicine
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Phase 2 Multicenter Clinical Trial of Intraoperative Molecular Imaging of Lung Cancer with a pH-Activatable Nanoprobe — https://pubmed.ncbi.nlm.nih.gov/38992245/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for surgical excision of pulmonary lesions were eligible for enrollment. The study was conducted at two large cancer surgical centers from from April 13, 2022 through August 31, 2022. Four patients withdrew consent prior to dosing.
Period: Overall Study
Arm/Group | Fluorescence Imaging With Pegsitacianine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Experiencing at Least One Clinically Significant Event (CSE)
Description: Discovery of a clinically significant event at the level of the patient. May include detection of primary tumors, discovery of occult disease, or tumor negative SOC biopsies.
Time Frame: 1 day
Population: Patients that received at least 75% of planned dose, had at least 1 image collected, and had disease present
Measure: Count of Participants; unit: Participants
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 16
Participants | 2

2. Secondary Outcome: Sensitivity of Pegsitacianine at Detecting Presence of Tumor Within the Tissue Specimen
Description: # of true positive specimens divided by the (#of true positive specimens + # of false negative specimens)
Time Frame: 7 days
Population: non-lymph node tissue specimens from lung resection
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 20
Number analyzed (tissue specimens) | 22
ratio | .32 [.125 to .566]

3. Secondary Outcome: Specificity of Pegsitacianine at Detecting Presence of Tumor Within the Tissue Specimen
Description: # of True Negative Specimens divided by the (# of True Negative Specimens + # of False Positive Specimens)
Time Frame: 7 days
Population: non-lymph node lung tissue specimens
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 20
Number analyzed (tissue specimens) | 22
ratio | .33 [.008 to .708]

4. Secondary Outcome: Negative Predictive Value of Pegsitacianine
Description: # of True negative specimens divided by the (# of true negative specimens + # of false negative specimens)
Time Frame: 7 days
Population: non-lymph node tissue specimens
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 20
Number analyzed (tissue specimens) | 22
ratio | .071 [.002 to .339]

5. Secondary Outcome: Positive Predictive Value of Pegsitacianine
Description: # of true positive specimens divided by the (# of true positive + # of false positive specimens)
Time Frame: 7 days
Population: non-lymph node lung tissue specimens
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 20
Number analyzed (tissue specimens) | 22
ratio | .75 [.349 to .968]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of infusion (24 hours prior to surgery) through 28 days post surgery.
Arm/Group | Fluorescence Imaging With Pegsitacianine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorescence Imaging With Pegsitacianine (N=20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — non-drug related complication due to surgical procedure
Subcutaneoius Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorescence Imaging With Pegsitacianine (N=20)
Procedural Pain (Injury, poisoning and procedural complications) | 16 (16)
Infusion Related Reactions (Injury, poisoning and procedural complications) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05048082/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT05048082/SAP_003.pdf